CLINICAL TRIAL: NCT04975282
Title: The Effects of Oral Feeding Methods in Preterm Infants on Transition to Full Breastfeeding and Discharge Time: A Retrospective Study
Brief Title: Comparison of Bottle and Cup Feeding on Transition to Full Breastfeeding and Discharge Time
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Zühal Çamur, Principal Investigator RN, PhD, Pamukkale University
Other Study IDs: Cup feeding, Bottle feeding
Record Dates: First submitted 2021-07-12; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Preterm; Feeding, Bottle; Feeding Behavior; Feeding, Breast
Keywords: Preterm infants; Bottle feeding; Cup feeding; Feeding methods; Breastfeeding
MeSH Terms: conditions — Premature Birth; Bottle Feeding; Feeding Behavior; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bottle Feeding: The bottle feeding method was being used in the NICU (1 January -31 December 2018).
  Interventions: Device: Bottle feeding
- Cup Feeding: The cup feeding method was being used in the NICU (1 January -31 December 2019).
  Interventions: Device: Cup feeding

INTERVENTIONS:
Device: Bottle feeding — Bottle was used as an alternative oral feeding method for preterm infants.
  Groups: Bottle Feeding
Device: Cup feeding — Cup was used as an alternative oral feeding method for preterm infants.
  Groups: Cup Feeding

SUMMARY:
Breastfeeding is the ideal feeding method and that in the absence of breastfeeding the bottle and cup feeding are common alternatives. There is a lack of evidence regarding superiority of either of these methods. This study aimed to evaluate bottle feeding and cup feeding in preterm infants on the outcomes of full breastfeeding and discharge time.

DETAILED DESCRIPTION:
An estimated 20 million infants are born preterm each year (>37 weeks) and this number is increasing. The preterm newborn population is potentially unable to be fed orally for a long time in the postnatal period.However, it is not a disease that preterm infants cannot be fed orally as soon as they are born. Since the physiological functions are not yet fully mature, their adaptation to the external uterine environment is more complicated.This situation also means a long hospital stay. Therefore, the American Academy of Pediatrics (AAP) has determined oral feeding of the preterm baby as the main criterion for discharge.

In preterm infants, sucking and swallowing coordination occurs in the 32 to 34 gestation weeks.Oral feeding skills are developed by applying various sensorimotor interventions and cue-based feeding protocols to increase oral feeding performance.Tube feeding (orogastric and nasogastric) is widely preferred as their oral-motor skills are still immature.As postnatal age increases, alternative oral feeding methods are often used along with tube feeding.Bottle feeding, cup feeding spoon feeding and syringe feeding are the most popular methods in clinical practice. While determining the most available method of oral feeding in preterm infants, the selection criteria include their capacity to facilitate the transition to full breastfeeding to help sustain breastfeeding to shorten the duration of hospitalization and to ensure sufficient nutrition.

Direct full breastfeeding is the important and most recommended feeding method in new-borns. However, since full breastfeeding is not immediately possible in preterm infants, they definitely need an alternative feeding method.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (30-34 weeks);
* Considered medically stable
* With no facial deformity,
* Absent of neurological or congenital anomalies,
* Did not require sedation or vasoactive drugs
* Mother is providing breast milk & plans to breastfeed.

Exclusion Criteria:

* Presence of gastrointestinal conditions that complicate feeding such as NEC,
* Absence of mother,
* Absence of breast milk, and
* Preterm infants fed only formula

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants between 30-34 weeks and healthy
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Transition to Full Breastfeeding | From transition to breastfeeding, up to 1 week.
  Preterm infants fed with bottle (n=78) and cup (n=80) were compared in terms of transition to full breastfeeding. The transition period from oral feeding to full breastfeeding is different for every preterm infants. There is no specific time frame in the study. For this outcome, infants were evaluated for time from oral feeding to full breastfeeding.
Discharge Time | From admission to discharge, up to 4 weeks
  Preterm infants fed with bottle (n=78) and cup (n=80) were compared in terms of discharge times. There is no specific time frame in the study. For this outcome, infants were evaluated for lenght of stay hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Zühal Çamur, RN, PhD, Principal Investigator — Pamukkale University; Bengü Çetinkaya, RN, PhD, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No